CLINICAL TRIAL: NCT04464993
Title: StandUPTV: Reducing Sedentary Screen Time in Adults
Acronym: StandUPTV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA239612 (NIH)
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Sedentary Behavior; Screen Time; Physical Activity; Sleep
Keywords: Multiphase optimization strategy; Mobile health
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Investigators will use the multiphase optimization (MOST) framework to conduct a highly efficient full-factorial experimental study to simultaneously test the main effects for each of three intervention components (LOCKOUT, TEXT, EARN) and their interactions (e.g., TEXT+EARN; LOCKOUT+EARN+TEXT) over 16 weeks.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not have access to study arm assignment and participants will be encouraged not to divulge their study arm assignment during assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- CORE (Experimental): Participants will receive a "core" intervention which will include a basic version of the StandUPTV app and a Fitbit watch to use throughout the 16-week intervention.The Fitbit will provide device-based behavioral feedback through the StandUPTV self-monitoring component. SST feedback will be Self-monitoring will provide passive and objective feedback regarding SST behaviors and MVPA drawn from Fitbit and SCREENTIME sources. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. As part of this education, all participants will be provided a behavioral target of reducing their SST by 50% from their baseline. This target will be customized for the participant within StandUPTV based on a baseline week of observation.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE
- CORE + text (Experimental): CORE components + The TEXT component uses app-based prompts (i.e., prompts generated through StandUPTV app) that will provide simple adaptive content based upon length of most recent SST bout and time of day. These prompts will specifically target outcome expectations around SST and MVPA.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Context-based prompts: TEXT
- CORE + Lockout (Experimental): CORE components + Lockout component will enforce a 50% per week reduction in SST, based upon a baseline week of observation. If SST reaches the prescribed threshold, the investigators will use the limits from the StandUPTV app to restrict screen time through the end of the week (Monday-Sunday); at which point, 50% baseline allotment will be reinstated for an additional week. Participants will be provided with a planning tool for planning SST on a daily basis in order to reach their over 50% reduction goal.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Sedentary Screen Time lockout: LOCKOUT
- CORE + Earn (Active Comparator): CORE components + the investigators will enforce a 50% per week reduction in SST, based upon a baseline week of observation. If SST reaches the prescribed threshold, the investigators will use the limits from the StandUPTV app to restrict screen time through the end of the week (Monday-Sunday); at which point, 50% baseline allotment will be reinstated for an additional week. Participants will be provided a planning tool for planning SST on a daily basis in order to reach their over 50% reduction goal.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Earn sedentary screen time through moderate-vigorous physical activity: EARN
- CORE + Text + Earn (Active Comparator): Intervention components will be delivered as described in simpler factorial conditions.
  App shows progress toward SST goal or if goal is exceeded. Can earn additional SST through exercise based on 3:1 ratio , simple adaptive content (by SST bout, time of day). Lockout component will enforce a 50% per week reduction in SST, based upon a baseline week of observation.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Context-based prompts: TEXT; Behavioral: Earn sedentary screen time through moderate-vigorous physical activity: EARN
- CORE + Text + Lockout (Active Comparator): Intervention components will be delivered as described in simpler factorial conditions, and...
  If exceeded, the limits feature will restrict screen time through the end of the week (Monday-Sunday) so cannot exceed limit. Simple adaptive content (by SST bout, time of day).
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Sedentary Screen Time lockout: LOCKOUT; Behavioral: Context-based prompts: TEXT
- CORE + Earn + Lockout (Active Comparator): Intervention components will be delivered as described in simpler factorial conditions, and...
  If exceeded, the limits feature will restrict screen time through the end of the week (Monday-Sunday) so cannot exceed limit. Can earn additional SST through exercise based on 3:1 ratio.
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Sedentary Screen Time lockout: LOCKOUT; Behavioral: Earn sedentary screen time through moderate-vigorous physical activity: EARN
- CORE + Earn + Lockout + Text (Active Comparator): Intervention components will be delivered as described in simpler factorial conditions, and...
  If exceeded, the limits feature will restrict screen time through the end of the week (Monday-Sunday) so cannot exceed limit. Can earn additional SST through exercise based on 3:1 ratio). Simple adaptive content (by SST bout, time of day).
  Interventions: Behavioral: Device-based feedback, self-monitoring, and education: CORE; Behavioral: Sedentary Screen Time lockout: LOCKOUT; Behavioral: Context-based prompts: TEXT; Behavioral: Earn sedentary screen time through moderate-vigorous physical activity: EARN

INTERVENTIONS:
Behavioral: Device-based feedback, self-monitoring, and education: CORE — Participants will receive a "core" intervention which will include a basic version of the StandUPTV app on an android tablet and a Fitbit to use throughout the 16-week intervention.t. SST feedback will be provided within the smartphone application. Self-monitoring will provide passive and objective feedback regarding SST behaviors. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. As part of this education, all participants will be provided a behavioral target of reducing their SST by 50% from their baseline. This target will be customized for the participant within StandUPTV based on a baseline week of observation.
Behavioral: Sedentary Screen Time lockout: LOCKOUT — Sedentary Screen Time lockout: LOCKOUT Sedentary Screen Time lockout: LOCKOUT The investigators will enforce a 50% per week reduction in SST, based upon a baseline week of observation. If SST reaches the prescribed threshold, the investigators will use the limits feature to restrict screen time through the end of the week (Monday-Sunday); at which point, 50% baseline allotment will be reinstated for an additional week. Participants will be prompted to plan for their screen time and provided modest allowances for exceeding their screen time in a given week.
  Arms: CORE + Earn + Lockout; CORE + Earn + Lockout + Text; CORE + Lockout; CORE + Text + Lockout
Behavioral: Context-based prompts: TEXT — The TEXT component uses app-based prompts (i.e., prompts generated through StandUPTV, not text message based) that will provide simple adaptive content. Content of the prompts will be educational (i.e., based on risks of sedentary screen time) and motivational (i.e., advice to reduce sedentary screen time).
  Arms: CORE + Earn + Lockout + Text; CORE + Text + Earn; CORE + Text + Lockout; CORE + text
Behavioral: Earn sedentary screen time through moderate-vigorous physical activity: EARN — Earn sedentary screen time through moderate-vigorous physical activity: EARN Participants assigned to the EARN component will earn SST by engaging in a >5 min continuous bout of exercise (as defined by Fitbit minutes >4 metabolic equivalents). They will earn SST on a 3:1 ratio up until they reach their baseline level of MVPA (5 mins of exercise earns 15 mins of SST). They will receive behavioral strategies to reduce screen time within the app (e.g., self-efficacy, barriers, exercising safely) and a planning tool for scheduling MVPA.
  Arms: CORE + Earn; CORE + Earn + Lockout; CORE + Earn + Lockout + Text; CORE + Text + Earn

SUMMARY:
The goal of this study is to develop an optimized intervention for reducing leisure sedentary screen time (SST) in middle-aged adults with overweight or obesity. Investigators will use the multiphase optimization (MOST) framework to conduct a highly efficient full-factorial experimental study to simultaneously test the main effects for each of three intervention components (LOCKOUT, TEXT, EARN) and their interactions (e.g., TEXT+EARN; LOCKOUT+EARN+TEXT) over 16 weeks.

DETAILED DESCRIPTION:
Primary Aim: To identify which component(s) from three components under consideration for inclusion in StandUPTV reduce SST by >60 min per day per day at 16 weeks. The three components tested will be: (a) LOCKOUT (no vs. yes); (b) TEXT (no vs. yes); and (c) EARN (no vs. yes). The investigators will use a highly efficient experimental strategy to detect effects of individual components as well as all two- and three-way interactions.

The secondary aim of this study is to examine how reductions in SST displace time into other active behaviors, i.e., light-intensity physical activity (LPA), moderate-to vigorous physical activity (MVPA) and activity type (e.g., housework, walking, exercise behaviors). The investigators will use both device-based (activPAL3c) and self-report (ACT24) measures to understand whether SST displacement can increase active behaviors, particularly MVPA.

ELIGIBILITY:
Inclusion Criteria:

* 23-64.90 years of age
* BMI≥25 kg/m2
* 3+ h/day of SST
* Insufficiently active
* Own an Apple or Android smartphone/tablet
* Access to internet at home or unlimited data plan
* Willing to download StandUPTV
* Able to read/understand English
* Willing to be randomized

Exclusion Criteria:

* Current smoker (more than once per week)
* Major life event (e.g., move out of study area, pregnant)
* MVPA contraindicated
* Occupation requires media use or high amounts of physical activity
* Drug abuse, major illness and/or psychological disorder

Ages: 23 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Buman, PhD, Principal Investigator — Arizona State University; Sarah Keadle, PhD, Principal Investigator — California Polytechnic University - San Luis Obispo
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - California Polytechnic University San Luis Obispo, San Luis Obispo, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasanaj K, Leonard KS, Sears DD, Yu F, Petrov ME, Keadle SK, Buman MP. Bidirectional associations of recreational sedentary screen time and 24-h behaviors: a dynamic cross-sectional multilevel model analysis. J Act Sedentary Sleep Behav. 2026 Feb 1. doi: 10.1186/s44167-026-00096-0. Online ahead of print. PMID 41622211
- [Derived] Keadle SK, Hasanaj K, Leonard KS, Fernandez A, Freid L, Weiss S, Legato M, Anand H, Hagobian TA, Phillips SM, Phelan S, Guastaferro K, Seltzer RGN, Buman MP. StandUPTV: a full-factorial optimization trial to reduce sedentary screen time among adults. Int J Behav Nutr Phys Act. 2025 Jun 13;22(1):77. doi: 10.1186/s12966-025-01771-2. PMID 40514642
- [Derived] Keadle S, Hasanaj K, Leonard-Corzo KS, Fernandez A, Freid L, Weiss S, Legato M, Anand H, Hagobian T, Phillips S, Phelan S, Guastaferro K, Seltzer R, Buman M. StandUPTV: A full-factorial optimization trial to reduce sedentary screen time among adults. Res Sq [Preprint]. 2025 Feb 24:rs.3.rs-5984168. doi: 10.21203/rs.3.rs-5984168/v1. PMID 40060037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data collection was scheduled to begin in July 2020 but was delayed until June 21, 2021 because of COVID-19. Specifically, we removed planned cardiovascular biomarker assessment, and the protocol was modified to conduct all assessments virtually, which opened recruitment to those outside the Phoenix, AZ and San Luis Obispo areas but delayed the start of the study. Enrollment continued until April 2023, and data collection was completed in September 2023.
Pre-assignment Details: The participants were required to have ≥4 days of measured screen time (i.e., verification from the study server that tablet and WeMo data were transmitted > 10 h/day) during the baseline period and were asked to repeat the baseline test if they had < 4 days recorded.
Groups:
- CORE: Participants will receive a "core" intervention which will include a basic version of the StandUPTV app and a Fitbit watch.The Fitbit will provide device-based behavioral feedback through the StandUPTV self-monitoring component. SST feedback will be Self-monitoring will provide passive and objective feedback regarding SST behaviors and MVPA drawn from Fitbit and SCREENTIME sources. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. As part of this education, all participants will be provided a behavioral target of reducing their SST by 50% from their baseline. This target will be customized for the participant within StandUPTV based on a baseline week of observation.
  Device-based feedback, self-monitoring, and education: CORE: Participants will receive a "core" intervention which will include a basic version of the StandUPTV app on an android tablet and a Fitbit to use throughout the 16-week intervention.t. SST feedback will be provided within the smartphone application. Self-monitoring will provide passive and objective feedback regarding SST behaviors. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. As part of this education, all participants will be provided a behavioral target of reducing their SST by 50% from their baseline. This target will be customized for the participant within StandUPTV based on a baseline week of observation.
- CORE + Lockout: CORE components + Lockout component will enforce a 50% per week reduction in SST, based upon a baseline week. If SST reaches the prescribed threshold, the StandUPTV app will restrict screen time through the end of the week (Monday-Sunday). Participants will be provided with a planning tool for planning SST.
  Device-based feedback, self-monitoring, and education: CORE: Participants will receive a "core" intervention which will include a basic version of the StandUPTV app on an android tablet and a Fitbit to use. SST feedback will be provided within the smartphone application. Self-monitoring will provide passive and objective feedback regarding SST behaviors. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. As part of this education, all participants will be provided a behavioral target of reducing their SST by 50% from their baseline. This target will be customized for the participant within StandUPTV based on a baseline week of observation.
  Sedentary Screen Time lockout: LOCKOUT The investigators will enforce a 50% per week reduction in SST, based upon a baseline week of observation. If SST reaches the prescribed threshold, the investigators will use the limits feature to restrict screen time through the end of the week (Monday-Sunday); at which point, 50% baseline allotment will be reinstated for an additional week.
- CORE + Earn: CORE components + 50% per week reduction in SST, based upon a baseline week. If SST reaches the prescribed threshold, the investigators will use the limits from the StandUPTV app to restrict screen time through the end of the week (Monday-Sunday). Participants will be provided a planning tool for planning SST on a daily basis in order to reach their over 50% reduction goal.
  Device-based feedback, self-monitoring, and education: CORE: Participants will receive a basic version of the StandUPTV app on an android tablet and a Fitbit to use throughout the 16-week intervention. SST feedback will be provided within the smartphone application. Self-monitoring will provide passive and objective feedback regarding SST behaviors. StandUPTV will also contain basic education including information on the risks of SST and tips for reducing SST. All participants will be provided a behavioral target of reducing their SST by 50% from their baseline.
  EARN: Earn sedentary screen time through moderate-vigorous physical activity: EARN Participants assigned to the EARN component will earn SST by engaging in a >5 min continuous bout of exercise (as defined by Fitbit minutes >4 metabolic equivalents). They will earn SST on a 3:1 ratio up until they reach their baseline level of MVPA (5 mins of exercise earns 15 mins of SST). They will receive behavioral strategies to reduce screen time within the app (e.g., self-efficacy, barriers, exercising safely) and a planning tool for scheduling MVPA.
Period: Overall Study
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Started | 11 | 13 | 14 | 16 | 15 | 15 | 10 | 16
Completed | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
Not Completed | 1 | 4 | 3 | 1 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text | Total
Number analyzed (Participants) | 11 | 13 | 14 | 16 | 15 | 15 | 10 | 16 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (10.6) | 45.5 (12.7) | 47.0 (10.5) | 42.9 (12.7) | 40.8 (12.2) | 42.7 (10.9) | 41.5 (12.7) | 42.0 (11.7) | 42.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 13 | 10 | 12 | 8 | 14 | 90
  Male | 1 | 2 | 2 | 3 | 5 | 3 | 2 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 3 | 2 | 3 | 2 | 3 | 23
  Not Hispanic or Latino | 9 | 8 | 11 | 13 | 13 | 12 | 8 | 13 | 87
  Unknown or Not Reported | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 9 | 11 | 13 | 12 | 9 | 10 | 7 | 11 | 82
  Race: Black | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 5
  Race: Asian | 1 | 0 | 0 | 4 | 3 | 2 | 1 | 3 | 14
  Race: Other | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 6
  Race: Unknown | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Sedentary Screen Time
Description: Minutes per day as measured by Stand UPTV app and activPAL
Time Frame: Baseline to 16 weeks
Population: Analyzed sample with multiple imputation.
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Number analyzed (Participants) | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
minutes per day | -88.2 [-147.7 to -28.8] | -60.1 [-113.0 to -7.2] | -102.7 [-161.5 to -43.8] | -118.1 [-163.0 to -73.1] | -17.0 [-63.6 to 29.6] | -72.8 [-122.9 to -22.6] | -94.3 [-156.2 to -32.4] | -125.7 [-172.0 to -79.3]

2. Secondary Outcome: Changes in Moderate to Vigorous Physical Activity
Description: Changes in moderate to vigorous physical activity (minutes per day as measured by activPAL)
Time Frame: Baseline to16 weeks
Population: Analyzed sample with multiple imputation.
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Number analyzed (Participants) | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
minutes per day | -7.2 [-14.8 to 0.4] | -0.1 [-7.2 to 6.9] | 1.0 [-6.2 to 8.2] | -0.7 [-6.7 to 5.2] | 1.2 [-4.9 to 7.3] | -15.6 [-22.4 to -8.8] | 1.5 [-7.6 to 10.6] | 0.3 [-5.8 to 6.3]

3. Secondary Outcome: Changes in Time Spent Sitting
Description: Changes in time spent sitting (Minutes per day as measured by activPAL)
Time Frame: Baseline to 16 weeks
Population: Analyzed sample with multiple imputation.
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Number analyzed (Participants) | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
minutes per day | -29.7 [-84.5 to 25.1] | -38.6 [-87.4 to 103] | 27.9 [-22.9 to 78.7] | -8.2 [-49.2 to 32.8] | -14.9 [-58.2 to 28.4] | 1.5 [-45.2 to 48.3] | 56.4 [-4.8 to 117.5] | 2.1 [-40.0 to 44.3]

4. Secondary Outcome: Changes in Time Spent Standing
Description: Changes in minutes per day of standing time as measured by activPAL
Time Frame: Baseline and 16 weeks
Population: Analyzed sample with imputation
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Number analyzed (Participants) | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
minutes per day | -0.4 [-38.4 to 37.7] | 27.4 [-8.9 to 63.7] | -15.7 [-49.8 to 18.5] | -8.7 [-37.6 to 20.3] | 10.3 [-19.9 to 40.6] | -2.8 [-38.2 to 32.5] | -37.7 [-83.7 to 8.3] | 7.0 [-22.7 to 36.6]

5. Secondary Outcome: Changes in Time Spent Stepping
Description: Minutes per day as measured by activPAL
Time Frame: Baseline to 16 weeks
Population: Analyzed sample with imputation
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
Number analyzed (Participants) | 10 | 9 | 11 | 15 | 14 | 13 | 7 | 15
minutes per day | 0.9 [-18.8 to 20.7] | 3.3 [-13.2 to 19.8] | -0.2 [-16.7 to 16.4] | -3.1 [-16.4 to 10.3] | 5.9 [-8.3 to 20.1] | -12.0 [-28.4 to 4.5] | -4.3 [-23.4 to 14.8] | 4.4 [-9.5 to 18.3]

ADVERSE EVENTS:
Time Frame: Baseline to 16 weeks (end of intervention period).
Arm/Group | CORE | CORE + Text | CORE + Lockout | CORE + Earn | CORE + Text + Earn | CORE + Text + Lockout | CORE + Earn + Lockout | CORE + Earn + Lockout + Text
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/14 | 0/16 | 0/15 | 0/15 | 0/10 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/14 | 0/16 | 0/15 | 0/15 | 0/10 | 0/16
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/14 | 0/16 | 0/15 | 0/15 | 0/10 | 0/16

LIMITATIONS AND CAVEATS:
Owing to delays in initiating and slowing recruitment during the COVID-19 pandemic, we did not meet the enrollment targets. Trial concluded when funding ended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04464993/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT04464993/SAP_001.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT04464993/ICF_002.pdf